CLINICAL TRIAL: NCT02990234
Title: The Efficacy of Capsular Repair in Arthroscopic Femoroacetabular
Brief Title: Capsular Repair in FAI Impingement Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-2310
Record Dates: First submitted 2016-12-05; First posted 2016-12-13 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Hip Injuries
Keywords: Capsular Repair; FAI; Hip
MeSH Terms: conditions — Hip Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsular Repair (Active Comparator): Capsular Repair arm. The first hip is randomized, opposite treatment on second hip. One Hip will receive the capsular repair while the other hip will not.
  Interventions: Procedure: Capsular Repair
- No Capsular Repair (Placebo Comparator): Placebo arm. One hip is randomized to capsular repair while the other hip has no capsular repair.
  Interventions: Procedure: No Capsular Repair

INTERVENTIONS:
Procedure: Capsular Repair
  Arms: Capsular Repair
Procedure: No Capsular Repair
  Arms: No Capsular Repair

SUMMARY:
The Investigator's hypothesis is that capsular repair (after CAM or mixed Femoroacetabular Impingement (FAI) surgery) requiring moderate capsulotomy, would result in similar patient outcomes in the short, mid and long term, both clinically and radiographically, compared to those without capsular repair. The objective of this clinical trial is to evaluate the clinical efficacy with regards to pain, range of motion and return to work and activities of daily living. Secondary objective is to evaluate radiographic characteristics between both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 16-51 years of age.
2. Healthy patients undergoing hip arthroscopy due to Cam or mixed FAI
3. No major osteoarthritic (OA) changes according to X-Ray and surgery observation (Tonnis 0-1)
4. No previous hip surgery
5. No other influential disabilities in lower limbs
6. No chronic use of NSAID, analgesics, steroids or chemotherapy drugs
7. Base line activity level (Tegner 3 and above)

Exclusion Criteria:

1. Patients with concomitant disease that may affect joints
2. Patients with major ligamentous laxity
3. Patients who have undergone only minor vertical capsulotomy (as in small pincer only lesions)
4. Patients with extreme range of motion needs (such as ballet dancers)
5. Patients suffering from connective tissue disease
6. Patients suffering from bilateral symptomatic FAI that are being operated on for their first hip
7. Patients with relative or proven dysplastic hip determined by center edge angle and/or extreme version abnormalities as measured on apical CT/MR cuts and pelvic XR
8. Patients who needed Ilio-Psoas release
9. Patients whose cartilage hip status was defined as advanced OA during surgery
10. Patients who following surgery would be instructed to avoid full weight bearing on the operated hip for more than 4 weeks
11. Concomitant use of PRP (platelet rich plasma) or hyaluronic acid during the surgical procedure
12. Patients with preoperative hip stiffness

Ages: 16 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in iHOT Version 12 | Baseline, 6weeks, 12weeks, 6months, 1Year, 2Years

OTHER OUTCOMES:
Change in Marx activity score | Baseline, 6weeks, 12weeks, 6months, 1Year, 2Years
Change in Range of Motion | Baseline, 14days, 6weeks, 12weeks, 6months, 1Year, 2Years
Change in X-rays | 6weeks, 6months, 1Year
  XR will be used for initial evaluation and for post op resection assessment and long-term OA changes. X-rays will be done post-operatively at 6 weeks, 6 months and 1 year time-frames. All these x-rays are normally performed as standard of care.
Change in MRI | 6weeks, 6months
  MRI will be conducted at 6 weeks and 6 months post op to evaluate capsular healing status (primary radiological outcome measure), intra articular adhesions, extra articular scarring, labrum/cartilage status and resection assessment. This MRI will be paid by department funds.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mei-Dan, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bowman KF Jr, Fox J, Sekiya JK. A clinically relevant review of hip biomechanics. Arthroscopy. 2010 Aug;26(8):1118-29. doi: 10.1016/j.arthro.2010.01.027. PMID 20678712
- [Background] Byrd JW. Hip arthroscopy. J Am Acad Orthop Surg. 2006 Jul;14(7):433-44. doi: 10.5435/00124635-200607000-00006. No abstract available. PMID 16822891
- [Background] Philippon MJ, Schenker ML. Arthroscopy for the treatment of femoroacetabular impingement in the athlete. Clin Sports Med. 2006 Apr;25(2):299-308, ix. doi: 10.1016/j.csm.2005.12.006. PMID 16638493
- [Background] Kelly BT, Weiland DE, Schenker ML, Philippon MJ. Arthroscopic labral repair in the hip: surgical technique and review of the literature. Arthroscopy. 2005 Dec;21(12):1496-504. doi: 10.1016/j.arthro.2005.08.013. PMID 16376242
- [Background] Ranawat AS, McClincy M, Sekiya JK. Anterior dislocation of the hip after arthroscopy in a patient with capsular laxity of the hip. A case report. J Bone Joint Surg Am. 2009 Jan;91(1):192-7. doi: 10.2106/JBJS.G.01367. No abstract available. PMID 19122095
- [Background] Matsuda DK. Acute iatrogenic dislocation following hip impingement arthroscopic surgery. Arthroscopy. 2009 Apr;25(4):400-4. doi: 10.1016/j.arthro.2008.12.011. Epub 2009 Feb 1. PMID 19341927
- [Background] Benali Y, Katthagen BD. Hip subluxation as a complication of arthroscopic debridement. Arthroscopy. 2009 Apr;25(4):405-7. doi: 10.1016/j.arthro.2009.01.012. PMID 19341928
- [Background] Ilizaliturri VM Jr, Byrd JW, Sampson TG, Guanche CA, Philippon MJ, Kelly BT, Dienst M, Mardones R, Shonnard P, Larson CM. A geographic zone method to describe intra-articular pathology in hip arthroscopy: cadaveric study and preliminary report. Arthroscopy. 2008 May;24(5):534-9. doi: 10.1016/j.arthro.2007.11.019. Epub 2008 Feb 1. PMID 18442685